CLINICAL TRIAL: NCT05638217
Title: Prospective Cohort Study: Efficacy of the Use of 38% Silver Diamine Fluoride and 5% Sodium Fluoride Varnish in Patients 4 to 12 Years for the Treatment of Caries and Its Association With Other Aspects of Relevance
Brief Title: Efficacy of the Use of Silver Diamine Fluoride and Sodium Fluoride Varnish for the Treatment of Caries in Children
Status: Completed | Type: Observational
Sponsor: Universidad Mayor de San Simón (Other)
Collaborators: Universidad Privada del Valle, Sede Cochabamba (Unknown); Industria Química Farmacéutica SIGMA CORP S.R.L. Cochabamba, Bolivia (Unknown); NODK LLC, Oregón, EE. UU. (Unknown); Food Bank Bolivia (Unknown)
Responsible Party: Principal Investigator, Rodrigo Arce Cardozo, Associate Research Professor, Universidad Mayor de San Simón
Other Study IDs: DINV-CAV01-EC001
Record Dates: First submitted 2022-11-10; First posted 2022-12-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries in Children
Keywords: Oral Health; Dental Caries; Silver Diamine Fluoride; Caries in Children; CaviGuard®
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of 4 to 12 years old eligible to received dental cavity treatment: Patients of 4 to 12 years old that are eligible to received dental cavity treatment. The goal of this observational study is to identify the efficacy of silver diamine fluoride 38% followed by sodium fluoride varnish 5%, using "CaviGuard®" as delivery method, in a population with untreated dental caries age range 4 to 12 years old.
  Interventions: Combination Product: Silver diamine fluoride 38% followed by Sodium fluoride varnish 5%

INTERVENTIONS:
Combination Product: Silver diamine fluoride 38% followed by Sodium fluoride varnish 5% — 1)Completely drying of the affected area 2)10 microliters of silver diamine fluoride 38% (CaviGuard®) will be placed on the affected area 3)The affected area should be immediately covered with 20 microliters of fluoride varnish 5% (CaviGuard®) 4)Repeat steps 1-3 one or two more times for large caries at intervals of at least 2 days apart 5)Follow up evaluation of treatment success visits will be conducted at 6 and 12 months from the initial treatment.
  NOTE: This is a single intervention using the device registered as Caviguard® to apply both products (Silver diamine fluoride 38% followed by Sodium fluoride varnish 5% (®)) in sequence.
  Other Names: CaviGuard®, Silver Diamine Fluoride (SDF)

SUMMARY:
The goal of this observational study is to identify the efficacy of silver diamine fluoride 38% followed by sodium fluoride varnish 5% in a population with untreated dental caries age range 4 to 12 years old. The main questions to answer are

* Efficacy of treatment of active tooth decay with the treatment protocol of 38% silver diamine fluoride and 5% sodium fluoride varnish.
* Clinical evaluation of tooth decay treated with 38% silver diamine fluoride and 5% sodium fluoride varnish in quality of hardness, color change and caries progression.
* Explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with: i. Reduction of oral pain caused by the presence of carious lesions. ii. Improvement in gingival oral health. iii. Changes in general nutritional status through measurements of height, weight, hemoglobin levels and nutritional survey. The participants will be identified, charted (with nutritional surveys and parameters), as well as treated and compared in a six- and twelve-month period, where researchers will clinically identify the association between the use of this protocol and the efficacy of such, as well as other related nutritional aspects.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to receive all necessary treatments and may be followed up for additional treatments and/or record follow-ups at each time point and for the duration of the study.
* Children within the age range mentioned above.
* Require a completed informed consent form and completed nutritional survey record for anyone who will participate in the program.
* According to the evaluation of the dentist Caries grade I and grade II
* In the case of patients with disabilities, at least one parent or legal guardian must be present at all times during the study.

Exclusion Criteria:

* Patients who, after assessment, identify a pulp condition or abscess in any of the teeth, this affected piece will be excluded from receiving treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish (in these cases, the Patient Coordinator will refer to a dentist outside the study for their treatment)
* Patients with caries with grade III or grade IV
* Patients with a known allergy to any of the active ingredients ( 38% silver diamine fluoride and 5% sodium fluoride varnish)
* Patients who were unable to give their informed consent or complete the nutritional survey.
* Patients who cannot participate during the entire program (12 months).
* Patients with other oral treatments (Orthodontics).
* Patients who are not present with at least one parent or legal guardian at the time of treatment.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be carried out in the city of Cochabamba, Bolivia, specifically at the Bolivian Food Bank Foundation located on Calle Francisco Prada between Aurelio Melean and J. Arauco 1120, from November 2022 to November 2023. This is a prospective cohort with a single assignment group (children aged 4 to 12 years) where a sample of 100-150 patients will be evaluated before, during and after their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Ratio of arrested cavity lesions after treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish | 6 months from initial treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions arrested after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist conducting an evaluation of multiple clinical findings including signs and symptoms of an active or arrested cavity.The clinical evaluation will be recorded in an odontograph for each patient.
Ratio of arrested cavity lesions after treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish | 12 months from treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist conducting an evaluation of multiple clinical findings including signs and symptoms of an active or arrested cavity.The clinical evaluation will be recorded in an odontograph for each patient.

SECONDARY OUTCOMES:
Evaluate hardness | 6 months from treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include hardness. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable hardness.
Evaluate color change | 6 months from treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include color change.The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable color change.
Evaluate cavity progression of cavity treated | 6 months from treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include cavity progression.The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable cavity progression.
Evaluation the reduction of oral pain caused by the presence of carious lesions. | 6 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the reduction of oral pain caused by the presence of carious lesions. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable reduction of oral pain.
Evaluate Improvement in gingival oral health. | 6 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the Improvement in gingival oral health. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable gingival oral health.
Evaluate changes in height and weight | 6 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through measurements of height and weight that will be combined with height and weight for age in child grow standards from the world health organization.
Evaluate changes in hemoglobin levels | 6 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through measurements of hemoglobin levels recorded as (g/dl).
Evaluate changes in a nutritional survey | 6 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through a 59 question nutritional survey developed by the research team.
Evaluate hardness | 12 months from initial treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include hardness. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable hardness.
Evaluate color change | 12 months from initial treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include color change.The clinical evaluation will be recorded odontograph for each patient and include dichotomous variables (yes/no) for the variable color change.
Evaluate cavity progression of cavity treated | 12 months from initial treatment
  The investigators will evaluate the efficacy of treatment of active cavity lesions after using the treatment protocol with 38% silver diamine fluoride and 5% sodium fluoride varnish. This evaluation will be performed by a trained dentist, conducting an evaluation of clinical finding that include cavity progression.The clinical evaluation will be recorded odontograph for each patient and include dichotomous variables (yes/no) for the variable cavity progression.
Evaluation of the reduction of oral pain caused by the presence of carious lesions | 12 months from initial treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the reduction of oral pain caused by the presence of carious lesions. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable reduction of oral pain.
Evaluate Improvement in gingival oral health. | 12 months from initial treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the Improvement in gingival oral health. The clinical evaluation will be recorded in an odontograph for each patient and include dichotomous variables (yes/no) for the variable gingival oral health.
Evaluate changes in height and weight | 12 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through measurements of height and weight that will be combined with height and weight for age in child grow standards from the world health organization.
Evaluate changes in hemoglobin levels | 12 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through measurements of hemoglobin levels recorded as (g/dl).
Evaluate changes in a nutritional survey | 12 months from treatment
  The investigators will explore the association of treatment with 38% silver diamine fluoride and 5% sodium fluoride varnish with the patient nutritional status through a 59 question nutritional survey developed by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Campero Ferrufino, DDS, Principal Investigator — Private University of the Valley; Ximena Claros Martinez, DDS, Principal Investigator — Private University of the Valley; Edwin Guarayo Molina, DDS, Principal Investigator — Private University of the Valley; Rodrigo k Arce Cardozo, MD, MPH,, Principal Investigator — Universidad Mayor de San Simon; Steve Duffin, DDS, Principal Investigator — NODK LLC
Locations (1):
- Bolivian Food Bank Foundation, Cochabamba, Bolivia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Intervention — https://caviguard.com/
- See also: Private University of the Valley — http://www.univalle.edu/